CLINICAL TRIAL: NCT01652430
Title: Experiential Avoidance in Combat Veterans With and Without Posttraumatic Stress Disorder
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 10-0159
Record Dates: First submitted 2011-12-09; First posted 2012-07-30 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2012-07

CONDITIONS: PTSD; Suicidal Ideation
Keywords: PTSD; Suicidal ideation; Cognitive processes
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Suicidal Ideation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PTSD cohort
- No PTSD cohort

SUMMARY:
This study plans to examine if symptoms of PTSD affect how Veterans who have served in combat think and react to certain information, and whether or not this has an influence on suicidal thoughts.

ELIGIBILITY:
Inclusion Criteria:

1. History of combat service
2. Diagnosis of PTSD confirmed by the CAPS or
3. No current diagnosis of PTSD
4. Age 18-65

Exclusion Criteria:

1. Inability to adequately respond to questions regarding the informed consent procedure.
2. History of significant neurological disease
3. Diagnosis of Schizophrenia or other Psychosis
4. Alcohol abuse/dependence or illicit drug use in the two weeks prior to testing
5. No history of combat service

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample for the current project will be recruited from the group of veterans receiving or eligible to receive outpatient mental health services at the Denver VA Medical Center who have served in combat who may or may not have a diagnosis of PTSD.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2010-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Beck Scale for Suicidal ideation | One time

CONTACTS AND LOCATIONS:
Overall Officials: Nazanin Bahraini, Ph.D., Principal Investigator — VA Eastern Colorado Healthcare System/MIRECC
Locations (1):
- Denver VA Medical Center, Denver, Colorado, United States